CLINICAL TRIAL: NCT00458757
Title: The Effect of Upper Arm Amputation and the Use of Prosthetics on Spatial Visual Representation in Peripersonal Space - a Behavioural Study
Brief Title: The Effect of Amputation on Spatial Visual Representation in Peripersonal Space
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 090767-amputy-HMO-CTIL
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2007-03

CONDITIONS: Upper Limb Amputees
Keywords: Amputees; Affordance; Peripersonal space; Pseudo neglect; Reaching; Spatial; visual
MeSH Terms: conditions — Personal Space

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
In this study, we wish to find behavioral evidence for the question whether an amputation of the arm can lead to changes in visual perception or motor responses to objects in peripersonal space. We hypothesize that changes in the motor and somatosensory hand-related cortices following amputation might lead to changes in parietal hand-related areas. The consequence of these parietal changes should be reflected behaviorally in reduced perception/attention/responses to hand-related objects in the space ipsilateral to the amputation. We further hypothesize that the use of prosthetics may provide the necessary visual feedback to maintain an intact hand representation and therefore lead to lesser cortical reorganization in both visual and somatosensory cortical areas.

DETAILED DESCRIPTION:
In a recent fMRI study (Makin TR. et al., J. Neurosci. 2007), we found extended cortical representation for a visual stimulus provided that it is presented close to the hand. It is therefore interesting to ask whether changes in the brain following limb amputation might induce changes in the amputees' perception of the body and consequently it's surrounding. In this study, we wish to find behavioral evidence for the question whether an amputation of the arm can lead to changes in visual perception or motor responses to objects in peripersonal space. We hypothesize that changes in the motor and somatosensory hand-related cortices following amputation might lead to changes in parietal hand-related areas. Consequently, we expect to find reduced perception/attention/responses to hand-related objects in the space ipsilateral to the amputation.

In this experiment we plan to employ a paradigm which is inspired by the affordance effect, originally introduced by Tucker and Elice (1998): we will present subjects with brief images of either manipulable or non manipulable objects in either the left or right visual field. The subjects will be required to determine whether the object contains a metal or not, by moving either their left or their right shoulder. We predict that while the control group of normal subjects would show a congruency effect (that is superior performance (faster and more accurate responses) when the responding shoulder is congruent with the position of the objects, the amputees will show spatial biases towards the non-amputated side. This effect should be more prominent for the manipulable objects.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb amputee, amputation above wrist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this experiment we plan to employ a paradigm which is inspired by the affordance effect, originally introduced by Tucker and Elice (1998): we will present subjects with brief images of either manipulable or non manipulable objects in either the left or right visual field. The subjects will be required to determine whether the object contains a metal or not, by moving either their left or their right shoulder. We predict that while the control group of normal subjects would show a congruency effect (that is superior performance (faster and more accurate responses) when the responding shoulder is congruent with the position of the objects, the amputees will show spatial biases towards the non-amputated side. This effect should be more prominent for the manipulable objects.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-11

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Schuartz, MD, Principal Investigator — Rehabilitation Dep. Hadassah Medical Hospital, Mount Scopus, Jerusalem
Locations (1):
- Neurobiology Dep., Life Sciences Institute, Hebrew Uni., Jerusalem, Israel

REFERENCES:
- [Background] Makin TR, Holmes NP, Zohary E. Is that near my hand? Multisensory representation of peripersonal space in human intraparietal sulcus. J Neurosci. 2007 Jan 24;27(4):731-40. doi: 10.1523/JNEUROSCI.3653-06.2007. PMID 17251412
- [Background] Tucker M, Ellis R. On the relations between seen objects and components of potential actions. J Exp Psychol Hum Percept Perform. 1998 Jun;24(3):830-46. doi: 10.1037//0096-1523.24.3.830. PMID 9627419